CLINICAL TRIAL: NCT04310956
Title: A Multi-center, Randomized Controlled Trial to Evaluate the Effectiveness and Safety of Y-Knot All-suture Anchor in Ankle Ligaments Injury Repair
Brief Title: A RCT for Y-Knot All-suture Anchor in Ankle Ligaments Injury Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ConMed Linvatec Beijing (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P18101
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2021-08

CONDITIONS: Ligament Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Y-Knot group (Experimental): Patients use Y-Knot all-suture anchor
  Interventions: Device: Y-Knot all-suture anchor
- Biocomposite suture anchor (Active Comparator): Patients use Biocomposite suture anchor
  Interventions: Device: Biocomposite suture anchor

INTERVENTIONS:
Device: Y-Knot all-suture anchor — Y-knot all-suture anchor will be implanted to participants
  Arms: Y-Knot group
Device: Biocomposite suture anchor — Biocomposite suture anchor will be implanted to participants
  Arms: Biocomposite suture anchor

SUMMARY:
Purpose of this study is to evaluate the effectiveness and safety of Y-Knot all-suture anchor by comparing patients' clinical outcome after ankle ligaments repair surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, no less than 18 years old;
* Patient was diagnosed as Collateral Ligament injury or Achilles tendon injury based on MRI or X-Ray who need to conduct foot&ankle repair surgery by investigator;
* Patient willing to sign a written consent form participating in this study；
* Subject is able to understand study, willing to comply the study procedures, and willing to return to hospital for follow-up up to 6 months postoperative；
* Life expectancy is more than 2 years post-operationally;

Exclusion Criteria:

* Conducted surgery at index ankle and possibly influence the outcome evaluation;
* Bilateral ankle surgery;
* Suffering concurrent ankle disease that may leads to a surgery during the study phase;
* known or suspected allergies to implant and/or instrument materials;
* pathological conditions of bone which would adversely affect the anchor fixation; with concurrent severe injury at index leg that may influence the outcome evaluation; Severe obesity;
* With concurrent disease that may influence the index ankle function;
* Patients with active sepsis or infection;
* With concurrent disease that may influence the stability of device and rehabilitation;
* Immune suppression, impairment of immune function, or autoimmune disease;
* Pregnant or lactating women;
* Known noncompliance or lost follow-up risk;
* Participated other drug, biologic, or device clinical trial 12 months before enrollment;
* Alcohol or drug abuser;
* Other inappropriate condition based on investigator determination;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
improvement of AOFAS score | From pre-operation to 6 months postoperative

SECONDARY OUTCOMES:
improvement of AOFAS score | From pre-operation to 3 months postoperative
Improvement of VAS score | From pre-operation to 3 and 6 months postoperative
ligament injury recurrences | up to 6 months postoperative
secondary surgery | up to 6 months postoperative

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Huashan Hosptial, Shanghai, Shanghai Municipality
  - Sichuan Orthopedics Hospital, Chengdu
  - Qilu Hospital of Shandong University, Jinan
  - Shenzhen Second People's Hospital, Shenzhen

IPD SHARING:
Plan to Share IPD: No